CLINICAL TRIAL: NCT03393806
Title: A Double Blind (Sponsor Open) Placebo-controlled, Stratified, Parallel Group Study to Evaluate the Efficacy and Safety of Repeat Doses of GSK3772847 in Participants With Moderate to Severe Asthma With Allergic Fungal Airway Disease (AFAD)
Brief Title: Repeat Dose Study of GSK3772847 in Participants With Moderate to Severe Asthma With Allergic Fungal Airway Disease (AFAD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was terminated early before meeting target enrolment due to a high screen failure rate and the feasibility of completing the study in a timely way
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207972; 2017-003544-20 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Asthma
Keywords: Asthma Control Questionnaire; Allergic fungal airway disease; Asthma Quality of Life Questionnaire; Holter monitoring; Asthma
MeSH Terms: conditions — Asthma | interventions — melrilimab

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either 10 mg/kg GSK3772847 or matching placebo intravenously.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving GSK3772847 (Experimental): Participants will be randomized to receive GSK3772847 as IV infusion. Participants will receive three doses ( Day 1, Day 29 and Day 57) of GSK3772847 every 4 weeks
  Interventions: Drug: GSK3772847
- Participants receiving placebo (Placebo Comparator): Participants will be randomized to receive matching placebo as IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3772847 — GSK3772847 will be available as 100 mg/vial, white to yellow, uniform lyophilized cake in a 5 milliliter (mL) clear glass vial with closure sealed by red metal and yellow overseal.
  Arms: Participants receiving GSK3772847
Drug: Placebo — Commercially sourced sterile normal saline will be provided as Placebo
  Arms: Participants receiving placebo

SUMMARY:
This study is multicenter, double-blinded parallel group design, where participants with moderate to severe asthma with AFAD will be enrolled. Participants will receive three doses of 10 milligrams/kilogram (mg/kg) of GSK3772847 every 4 Weeks versus placebo along with standard of care. Participants will be randomized in 1:1 ratio to receive either 10 mg/kg GSK3772847 intravenously (IV) or matching placebo IV. Participants will receive study treatment on Week 0 (Day 1), Week 4 and Week 8. The total duration of the study will be 28 Weeks and approximately 46 participants will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age inclusive, at the time of signing the informed consent.
* Documented history of physician diagnosed moderate or severe asthma for >=12 months based on Guidelines and treated with inhaled corticosteroid (ICS) and long-acting beta-2-agonist (LABA) for at least 4 months (>=500 micrograms/day [µg/day]) fluticasone propionate or equivalent as defined in the guidelines.
* Pre-bronchodilator FEV1 35-79% of predicted value for participant inclusive
* FeNO >= 25 parts per billion (ppb) at Screening
* ACQ-5 score >= 1.5 at Screening
* Blood eosinophil >=300 cells/microliter at Screening
* Evidence of allergic fungal airway disease like Fungal sensitization to any of the fungi Aspergillus fumigatus, Penicillium chrysogenum (notatum) at screening measured by serum-specific Immunoglobulin (Ig) E test. A history of exacerbations with at least 1 severe exacerbation (defined as requiring a minimum of 3 days of high-dose oral corticosteroids for asthma symptoms) in the previous 12 months.
* Body weight within 50-150 kilogram (kg)
* Both male and female gender. A female participant is eligible to participate if she is not pregnant not breastfeeding, Not a woman of childbearing potential (WOCBP) or A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 16 weeks after the last dose of study treatment.
* Capable of giving signed informed consent

Exclusion Criteria:

* Historical diagnosis of cystic fibrosis
* Concurrent respiratory diseases: Presence of a known pre-existing, clinically important respiratory conditions (example pneumonia, pneumothorax, atelectasis segmental or larger, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities) other than asthma or AFAD
* Has a history of chronic or recurrent non-pulmonary infectious disease or ongoing non-pulmonary infection including, but not limited to, chronic renal infection, chronic chest infection, recurrent urinary tract infection (example, recurrent pyelonephritis, chronic non-remitting cystitis), or open, draining skin wound or an ulcer
* Serious infection within 8 weeks of enrolment, including, but not limited to hepatitis, pneumonia, sepsis, or pyelonephritis; or has been hospitalized for an infection; or has been treated with IV antibiotics for an infection, within 8 weeks prior to the first administration of study drug.
* Evidence of poorly controlled chronic medical conditions other than asthma, example, participants with known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, cardiovascular, gastrointestinal, hepatic, and hematological or any other system abnormalities that are uncontrolled with standard treatment.
* Cardiovascular disease: Clinically significant organic heart disease
* Participants with a diagnosis of malignancy or in the process of investigation for a malignancy. Participants with carcinoma that have not been in complete remission for at least 5 years. Participants who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the participant has been considered cured by treatment.
* Eosinophilic diseases: Other conditions that could lead to elevated eosinophil such as hyper-eosinophilic syndromes. Participants with a known, pre-existing parasitic infestation within 6 months prior to Screening (Visit 1)
* Prohibited medications is not permitted within the defined time intervals prior to Screening (Visit 1) and throughout the study.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A known immunodeficiency such as human immunodeficiency virus infection.
* Hypersensitivity: significant allergies to humanized monoclonal antibodies or biologic or to any components of the formulation used in this study
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear Ig A dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Clinically significant abnormality on 12-lead ECG assessment at screening (Visit 1). Site investigators will be provided with ECG over-read conducted by a centralized independent cardiologist, to assist in evaluation of participant eligibility.
* Sinus bradycardia <45 beats per minute (bpm), sinus tachycardia >= 110 bpm, multifocal atrial tachycardia (wandering atrial pacemaker with rate >100bpm), evidence of Mobitz II second degree or third degree atrioventricular (AV) block, pathological Q waves (defined as wide [>0.04 seconds] and deep [>0.4 millivolts (mV) (4 millimeter [mm] with 10mm/mV setting)] or >25% of the height of the corresponding R wave, providing the R wave was >0.5mV [5mm with 10mm/mV setting], appearing in at least two contiguous leads, evidence of ventricular ectopic couplets, bigeminy, trigeminy or multifocal premature ventricular complexes, for participants without complete right bundle branch block: QTc for heart rate by Fridericia's formula QTc(F) >= 450 millisecond (msec) or an ECG that is unsuitable for QT measurements, for participants with complete right bundle branch block: QTc(F) >=480 msec or an ECG that is unsuitable for QT measurements, ST-T wave abnormalities, clinically significant conduction abnormalities and clinically significant arrhythmias.
* Smoking history: current smokers or former smokers with a smoking history >= 10 pack years
* History of alcohol or illegal substance abuse within 2 years prior to Screening (Visit1).
* Participants at risk of non-compliance, or unable to comply with the study procedures. Participants who are unable to follow study instructions such as visit schedule and paper diary completion. Participants who have known evidence of lack of adherence to controller medication and/or ability to follow physician's recommendations. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- France (3):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
- GSK Investigational Site, Amsterdam, Netherlands
- Russia (5):
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ulyanovsk
- United Kingdom (6):
  - GSK Investigational Site, Wythenshawe, Greater Manchester
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Edgbaston

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Akinseye C, Crim C, Newlands A, Fairman D. Efficacy and safety of GSK3772847 in participants with moderate-to-severe asthma with allergic fungal airway disease: A phase IIa randomized, multicenter, double-blind, sponsor-open, comparative trial. PLoS One. 2023 Feb 3;18(2):e0281205. doi: 10.1371/journal.pone.0281205. eCollection 2023. PMID 36735745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double-blind, placebo-controlled, parallel group study conducted in participants with moderate to severe asthma with allergic fungal airway disease (AFAD). The study was conducted across 4 countries-France, Netherlands, Russian Federation and the United Kingdom.
Pre-assignment Details: A total of 17 participants were randomized in a ratio of 1:1 to receive either GSK3772847 10 milligrams per kilogram (mg/kg) or placebo. Recruitment in the study was terminated early due to the feasibility of completing the study in a timely manner.
Groups:
- Placebo: Participants received three doses of placebo administered intravenously every 4 weeks (Weeks 0, 4 and 8) along with their standard of care treatment.
- GSK3772847: Participants received three doses of GSK3772847 10 mg/kg administered intravenously every 4 weeks (Weeks 0, 4 and 8) along with their standard of care treatment.
Period: Overall Study
Arm/Group | Placebo | GSK3772847
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3772847 | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (9.57) | 53.6 (12.59) | 56.9 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Japanese/East Asian (EA)/South EA Heritage | 0 | 2 | 2
  White | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Blood Eosinophils Over Time
Description: Blood samples were collected at the indicated time points for assessment of blood eosinophil cell count. Baseline is the most recent recorded value before dosing on Day 1. Percent change from Baseline is calculated as (Ratio to Baseline minus 1)*100, where ratio to Baseline is the value at specified time point divided by Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Weeks 2, 4, 8 and 12
Population: Modified Intent-to-Treat (mITT) Population comprised of all randomized participants who took at least 1 dose of study treatment. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Percent change
  Week 2; n=9, 8 | 30.8 [4 to 61] | 28.1 [-46 to 550]
  Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4; n=8, 8 | 16.0 [-17 to 77] | 2.1 [-71 to 469]
  Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8; n=8, 8 | 14.4 [-98 to 262] | -31.4 [-59 to 10]
  Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Week 12; n=5, 7 | 9.7 [-88 to 67] | -10.9 [-76 to 469]

2. Primary Outcome: Percent Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) Over Time
Description: FeNO was assessed using a handheld electronic device. The measurements were obtained in accordance with the American Thoracic Society and the European Respiratory Society Recommendations for Standardized Procedures for the Online and Offline Measurement of Exhaled Lower Respiratory Nitric Oxide and Nasal Nitric Oxide. Participants did not use their rescue medication for at least 6 hours before each FeNO assessment, unless essential for clinical need. Baseline is the most recent recorded value before dosing on Day 1. Percent change from Baseline is calculated as (Ratio to Baseline minus 1)*100, where ratio to Baseline is the value at specified time point divided by Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Weeks 2, 4, 8 and 12
Population: mITT Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Percent change
  Week 2; n=9, 6: number analyzed (Participants) | 9 | 6
  Week 2; n=9, 6 | 33.4 [-39 to 51] | -18.6 [-37 to 12]
  Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4; n=8, 8 | 13.7 [-29 to 205] | -12.5 [-48 to 36]
  Week 8; n=8, 7: number analyzed (Participants) | 8 | 7
  Week 8; n=8, 7 | 11.7 [-80 to 75] | -42.8 [-67 to 5]
  Week 12; n=5, 6: number analyzed (Participants) | 5 | 6
  Week 12; n=5, 6 | -37.2 [-65 to -16] | -45.6 [-68 to -34]

3. Secondary Outcome: Serum Concentrations of GSK3772847
Description: Whole blood samples were collected at indicated time points for measurement of serum concentrations of GSK3772847.
Time Frame: Week 0 (post-dose), Week 2, Week 4 (pre-dose), Week 8 (pre-dose and post-dose), Week 12 and Week 24
Population: Pharmacokinetic (PK) Population comprised of all randomized participants who received at least one dose of study medication, and for whom at least one pharmacokinetic sample was obtained, analyzed and was measurable.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | GSK3772847
Number analyzed (Participants) | 8
Micrograms per milliliter
  Week 0, post-dose | 156.50 (74.102)
  Week 2 | 65.35 (10.900)
  Week 4, pre-dose | 39.13 (10.777)
  Week 8, pre-dose | 56.24 (9.658)
  Week 8, post-dose | 209.61 (93.217)
  Week 12 | 68.59 (15.570)
  Week 24 | 1.67 (1.276)

4. Secondary Outcome: Serum Levels of Free Suppressor of Tumorigenicity 2 (ST2)
Description: Serum samples were collected at indicated time points for assessment of free ST2 levels. Baseline is the most recent recorded value before dosing on Day 1 (Week 0).
Time Frame: Baseline, Week 0 (post-dose), Week 2, Week 4 (pre-dose), Week 8 (pre-dose and post-dose) and Week 12
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Micrograms per liter
  Baseline; n=9, 8 | 2.365 (54.3) | 2.418 (50.0)
  Week 0 (post-dose); n=9, 8 | 2.301 (46.9) | 0.025 (668.2)
  Week 2; n=9, 8 | 2.286 (50.2) | 0.156 (43.4)
  Week 4 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4 (pre-dose); n=8, 8 | 2.382 (32.1) | 0.197 (44.0)
  Week 8 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8 (pre-dose); n=8, 8 | 2.563 (30.8) | 0.181 (25.8)
  Week 8 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8 (post-dose); n=8, 8 | 2.568 (33.7) | 0.126 (38.2)
  Week 12; n=5, 6: number analyzed (Participants) | 5 | 6
  Week 12; n=5, 6 | 2.194 (46.5) | 0.144 (67.3)

5. Secondary Outcome: Serum Levels of Total Soluble ST2
Description: Serum samples were collected at indicated time points for assessment of total soluble ST2 levels. Baseline is the most recent recorded value before dosing on Day 1 (Week 0).
Time Frame: Baseline, Week 0 (post-dose), Week 2, Week 4 (pre-dose), Week 8 (pre-dose and post-dose) and Week 12
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Micrograms per liter
  Baseline; n=9, 8 | 1.905 (71.4) | 2.382 (51.1)
  Week 0 (post-dose); n=9, 8 | 1.884 (60.4) | 3.258 (39.6)
  Week 2; n=9, 8 | 1.777 (65.5) | 63.353 (44.7)
  Week 4 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4 (pre-dose); n=8, 8 | 1.950 (35.6) | 65.833 (47.3)
  Week 8 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8 (pre-dose); n=8, 8 | 2.141 (39.9) | 79.286 (31.6)
  Week 8 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8 (post-dose); n=8, 8 | 2.201 (40.7) | 74.046 (44.7)
  Week 12; n=5, 6: number analyzed (Participants) | 5 | 6
  Week 12; n=5, 6 | 1.900 (61.3) | 75.703 (54.1)

6. Secondary Outcome: Number of Participants With Positive Anti-GSK3772847 Antibodies Post-dosing
Description: Serum samples were collected at indicated time points and tested for the presence of antibodies that bind to GSK3772847. The presence of anti-GSK3772847 antibodies was assessed using a tiered approach including a screening assay, a confirmation assay and calculation of titre. Data for participants who showed positive results for confirmation assay has been presented.
Time Frame: Weeks 0, 2, 4, 8, 12 and 24
Population: Safety Population consisted of all randomized participants who took at least 1 dose of study treatment. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Participants
  Week 0; n=9, 8 | 0 | 0
  Week 2; n=9, 8 | 0 | 0
  Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4; n=8, 8 | 0 | 0
  Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8; n=8, 8 | 0 | 0
  Week 12; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 12; n=8, 8 | 0 | 0
  Week 24; n=9, 8 | 0 | 0

7. Secondary Outcome: Number of Participants for Whom Titers of Anti-GSK3772847 Antibodies Was Performed
Description: Serum samples were collected at indicated time points and tested for the presence of antibodies that bind to GSK3772847. The presence of anti-GSK3772847 antibodies was assessed using a tiered approach including a screening assay, a confirmation assay and calculation of titer. Data for number of participants for whom titers of anti-GSK3772847 antibodies was performed is presented.
Time Frame: Weeks 0, 2, 4, 8, 12 and 24
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Participants
  Week 0; n=9, 8 | 0 | 0
  Week 2; n=9, 8 | 0 | 0
  Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4; n=8, 8 | 0 | 0
  Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8; n=8, 8 | 0 | 0
  Week 12; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 12; n=8, 8 | 0 | 0
  Week 24; n=9, 8 | 0 | 0

8. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Absolute Score at Weeks 2, 4, 8 and 12
Description: The ACQ-5 is a five-item, self-completed questionnaire, which measures a participant's asthma control. The questions enquire about the frequency and/or severity of symptoms (nocturnal awakening, activity limitation, shortness of breath and wheeze) over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/limitation) scale. ACQ-5 score is the mean of the five questions and ranges from 0 (totally controlled) to 6 (severely uncontrolled). Baseline value is defined as the ACQ-5 assessment on Day 1. Change from Baseline is calculated as the post-dose value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Scores on a scale
  Week 2; n=9, 8 | -0.47 (0.616) | -0.65 (0.739)
  Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4; n=8, 8 | -0.23 (1.087) | -1.03 (0.897)
  Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8; n=8, 8 | -0.60 (0.986) | -1.23 (1.383)
  Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Week 12; n=5, 7 | -0.12 (1.262) | -1.20 (1.095)

9. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Total and Domain Scores at Weeks 2, 4, 8 and 12
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire that was developed to evaluate the impact of asthma treatments on the quality of life of asthma sufferers. The AQLQ contains 32 items in four domains: activity limitation (11 items), symptoms (12 items), emotional function (five items), and environmental stimuli (four items). Participants were asked to recall their experience over the previous 14 days and respond to each question on a seven-point scale where a value of 1 indicates 'total impairment' and 7 indicates 'no impairment'. The total score is the mean of responses to all 32 questions and each individual domain score was calculated as the mean of the items within that domain. Hence, the total and domain scores were each defined on a range from 1 to 7 with higher scores indicating a higher quality of life. Baseline value is defined as the AQLQ assessment on Day 1. Change from Baseline is calculated as the post-dose value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Scores on a scale
  Total score: Week 2; n=9, 8 | 0.31 (0.660) | 0.45 (0.623)
  Total score: Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Total score: Week 4; n=8, 8 | -0.22 (0.477) | 0.56 (0.514)
  Total score: Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Total score: Week 8; n=8, 8 | 0.27 (0.846) | 1.09 (0.940)
  Total score: Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Total score: Week 12; n=5, 7 | 0.10 (1.394) | 1.13 (0.953)
  Activity limitation; Week 2; n=9, 8 | 0.20 (0.504) | 0.31 (0.750)
  Activity limitation; Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Activity limitation; Week 4; n=8, 8 | -0.26 (0.499) | 0.30 (0.570)
  Activity limitation; Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Activity limitation; Week 8; n=8, 8 | 0.12 (0.603) | 0.88 (0.900)
  Activity limitation; Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Activity limitation; Week 12; n=5, 7 | -0.07 (1.127) | 0.91 (0.993)
  Symptoms; Week 2; n=9, 8 | 0.52 (0.924) | 0.54 (0.641)
  Symptoms; Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Symptoms; Week 4; n=8, 8 | -0.05 (0.774) | 0.74 (0.627)
  Symptoms; Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Symptoms; Week 8; n=8, 8 | 0.57 (1.213) | 1.24 (0.936)
  Symptoms; Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Symptoms; Week 12; n=5, 7 | 0.52 (1.740) | 1.31 (0.810)
  Environmental stimuli; Week 2; n=9, 8 | -0.14 (0.811) | 0.22 (0.891)
  Environmental stimuli; Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Environmental stimuli; Week 4; n=8, 8 | -0.44 (0.884) | 0.63 (0.886)
  Environmental stimuli; Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Environmental stimuli; Week 8; n=8, 8 | -0.44 (1.208) | 1.06 (1.132)
  Environmental stimuli; Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Environmental stimuli; Week 12; n=5, 7 | -0.65 (1.025) | 0.89 (1.257)
  Emotional function; Week 2; n=9, 8 | 0.40 (0.860) | 0.75 (0.955)
  Emotional function; Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Emotional function; Week 4; n=8, 8 | -0.35 (0.833) | 0.65 (0.847)
  Emotional function; Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Emotional function; Week 8; n=8, 8 | 0.45 (1.165) | 1.22 (1.289)
  Emotional function; Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Emotional function; Week 12; n=5, 7 | 0.08 (1.712) | 1.37 (1.246)

10. Secondary Outcome: Percentage of Responders to ACQ-5 at Weeks 2, 4, 8 and 12
Description: The ACQ-5 is a five-item, self-completed questionnaire, which measures a participant's asthma control. The questions enquire about the frequency and/or severity of symptoms (nocturnal awakening, activity limitation, shortness of breath and wheeze) over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/limitation) scale. ACQ-5 score is the mean of the five questions and ranges from 0 (totally controlled) to 6 (severely uncontrolled). A responder to ACQ-5 is defined as a participant who has a decrease from Baseline in ACQ-5 score of 0.5 or more at Weeks 2, 4, 8 and 12.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Percentage of responders
  Week 2; n=9, 8 | 44 | 50
  Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4; n=8, 8 | 63 | 50
  Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8; n=8, 8 | 50 | 50
  Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Week 12; n=5, 7 | 20 | 71

11. Secondary Outcome: Percentage of Responders to AQLQ at Weeks 2, 4, 8 and 12
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire that was developed to evaluate the impact of asthma treatments on the quality of life of asthma sufferers. The AQLQ contains 32 items in four domains: activity limitation (11 items), symptoms (12 items), emotional function (five items), and environmental stimuli (four items). Participants were asked to recall their experience over the previous 14 days and respond to each question on a seven-point scale where a value of 1 indicates 'total impairment' and 7 indicates 'no impairment'. The total score is the mean of responses to all 32 questions. The total score was defined on a range from 1 to 7 with higher scores indicating a higher quality of life. A responder to AQLQ is defined as a participant who has an increase from Baseline in AQLQ score of 0.5 or more at Weeks 2, 4, 8 and 12.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Percentage of responders
  Week 2; n=9, 8 | 44 | 50
  Week 4; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4; n=8, 8 | 0 | 38
  Week 8; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8; n=8, 8 | 25 | 63
  Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Week 12; n=5, 7 | 40 | 86

12. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 is measured using spirometry. Baseline is the most recent recorded value before dosing on Day 1. Change from Baseline is calculated as the post-dose value minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Liters
  Week 2; n=9, 8 | 0.076 (0.3383) | -0.137 (0.2640)
  Week 4; n=7, 8: number analyzed (Participants) | 7 | 8
  Week 4; n=7, 8 | -0.049 (0.2304) | -0.022 (0.2703)
  Week 8; n=7, 7: number analyzed (Participants) | 7 | 7
  Week 8; n=7, 7 | 0.060 (0.4210) | 0.040 (0.2381)
  Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Week 12; n=5, 7 | 0.102 (0.4879) | -0.013 (0.1923)

13. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: FVC is the maximal amount of air that can be forcibly exhaled from lungs after taking the deepest breath possible. FVC is measured by spirometry. Baseline is the most recent recorded value before dosing on Day 1. Change from Baseline is calculated as the post-dose value minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Liters
  Week 2; n=9, 8 | 0.078 (0.4201) | -0.074 (0.3761)
  Week 4; n=7, 8: number analyzed (Participants) | 7 | 8
  Week 4; n=7, 8 | 0.091 (0.3163) | 0.090 (0.3049)
  Week 8; n=7, 7: number analyzed (Participants) | 7 | 7
  Week 8; n=7, 7 | 0.179 (0.5145) | 0.030 (0.2291)
  Week 12; n=5, 7: number analyzed (Participants) | 5 | 7
  Week 12; n=5, 7 | 0.136 (0.5351) | 0.050 (0.2408)

14. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Participants
  AEs | 7 | 3
  SAEs | 1 | 0

15. Secondary Outcome: Number of Participants With Worst Case Post-Baseline Chemistry Results Relative to Normal Range at Baseline
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, calcium, carbon dioxide, chloride, creatine kinase, creatinine, direct bilirubin, gamma glutamyl transferase, glucose, phosphate, potassium, protein, sodium and urea. Participants were counted in the worst case category that their value changed to (low, normal or high), unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent (%). 'To Low' rows are not presented for tests that have lower limit of normal = 0.
Time Frame: Up to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Participants
  Alanine aminotransferase; To normal or no change | 9 | 8
  Alanine aminotransferase; To high | 0 | 0
  Albumin; To low | 0 | 0
  Albumin; To normal or no change | 9 | 8
  Albumin; To high | 0 | 0
  Alkaline Phosphatase; To low | 0 | 0
  Alkaline Phosphatase; To normal or no change | 9 | 8
  Alkaline Phosphatase; To high | 0 | 0
  Aspartate Aminotransferase; To normal or no change | 9 | 8
  Aspartate Aminotransferase; To high | 0 | 0
  Bilirubin; To normal or no change | 9 | 8
  Bilirubin; To high | 0 | 0
  Calcium; To low | 0 | 1
  Calcium; To normal or no change | 9 | 7
  Calcium; To high | 0 | 0
  Carbon Dioxide; To low | 2 | 1
  Carbon Dioxide; To normal or no change | 7 | 7
  Carbon Dioxide; To high | 0 | 0
  Chloride; To low | 0 | 0
  Chloride; To normal or no change | 9 | 7
  Chloride; To high | 0 | 1
  Creatine Kinase; To normal or no change | 7 | 7
  Creatine Kinase; To high | 2 | 1
  Creatinine; To low | 0 | 1
  Creatinine; To normal or no change | 9 | 7
  Creatinine; To high | 0 | 0
  Direct Bilirubin; To normal or no change | 9 | 8
  Direct Bilirubin; To high | 0 | 0
  Gamma Glutamyl Transferase; To normal or no change | 9 | 8
  Gamma Glutamyl Transferase; To high | 0 | 0
  Glucose; To low | 0 | 0
  Glucose; To normal or no change | 7 | 7
  Glucose; To high | 2 | 1
  Phosphate; To low | 2 | 0
  Phosphate; To normal or no change | 5 | 8
  Phosphate; To high | 2 | 0
  Potassium; To low | 0 | 0
  Potassium; To normal or no change | 9 | 7
  Potassium; To high | 0 | 1
  Protein; To low | 0 | 1
  Protein; To normal or no change | 9 | 7
  Protein; To high | 0 | 0
  Sodium; To low | 0 | 0
  Sodium; To normal or no change | 8 | 7
  Sodium; To high | 1 | 1
  Urea; To low | 0 | 1
  Urea; To normal or no change | 9 | 7
  Urea; To high | 0 | 0

16. Secondary Outcome: Number of Participants With Worst Case Post-Baseline Hematology Results Relative to Normal Range at Baseline
Description: Blood samples were collected for the assessment of following hematology parameters: basophils, eosinophils, erythrocyte (Ery. ) mean hemoglobin concentration (MCHC), Ery. mean corpuscular hemoglobin (MCH), Ery mean corpuscular volume (MCV), erythrocytes, erythrocytes distribution width, hematocrit, hemoglobin, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Participants were counted in the worst case category that their value changed to (low, normal or high), unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. 'To Low' rows are not presented for tests that have lower limit of normal = 0.
Time Frame: Up to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Participants
  Basophils; To normal or no change | 9 | 8
  Basophils; To high | 0 | 0
  Eosinophils; To low | 1 | 0
  Eosinophils; To normal or no change | 5 | 6
  Eosinophils; To high | 3 | 2
  Ery. MCHC; To low | 4 | 0
  Ery. MCHC; To normal or no change | 5 | 8
  Ery. MCHC; To high | 0 | 0
  Ery. MCH; To low | 0 | 0
  Ery. MCH; To normal or no change | 9 | 8
  Ery. MCH; To high | 0 | 0
  Ery. MCV; To low | 0 | 0
  Ery. MCV; To normal or no change | 9 | 8
  Ery. MCV; To high | 0 | 0
  Erythrocytes; To low | 0 | 1
  Erythrocytes; To normal or no change | 9 | 7
  Erythrocytes; To high | 0 | 0
  EDW; To low | 0 | 0
  EDW; To normal or no change | 7 | 7
  EDW; To high | 2 | 1
  Hematocrit; To low | 1 | 1
  Hematocrit; To normal or no change | 8 | 6
  Hematocrit; To high | 0 | 1
  Hemoglobin; To low | 1 | 0
  Hemoglobin; To normal or no change | 8 | 8
  Hemoglobin; To high | 0 | 0
  Leukocytes; To low | 0 | 1
  Leukocytes; To normal or no change | 9 | 7
  Leukocytes; To high | 0 | 0
  Lymphocytes; To low | 0 | 0
  Lymphocytes To normal or no change | 9 | 8
  Lymphocytes; To high | 0 | 0
  Monocytes; To low | 1 | 2
  Monocytes; To normal or no change | 8 | 6
  Monocytes; To high | 0 | 0
  Neutrophils; To low | 1 | 1
  Neutrophils; To normal or no change | 7 | 7
  Neutrophils; To high | 1 | 0
  Platelets; To low | 0 | 0
  Platelets; To normal or no change | 9 | 8
  Platelets; To high | 0 | 0

17. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the supine position after five minutes of rest for the participant. Baseline is the most recent recorded value before dosing on Day 1 (Week 0). Change from Baseline is calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Week 0 (post-dose), Weeks 4 and 8 (pre-dose and post-dose) Weeks 12 and 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Millimeters of mercury
  SBP; Week 0 (post-dose); n=9, 8 | 3.7 (8.77) | 1.4 (9.38)
  SBP; Week 4 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  SBP; Week 4 (pre-dose); n=8, 8 | 0.1 (14.40) | -2.5 (18.05)
  SBP; Week 4 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  SBP; Week 4 (post-dose); n=8, 8 | 4.5 (14.16) | 4.5 (19.18)
  SBP; Week 8 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  SBP; Week 8 (pre-dose); n=8, 8 | 0.5 (14.42) | 7.3 (17.81)
  SBP; Week 8 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  SBP; Week 8 (post-dose); n=8, 8 | 0.6 (15.27) | 6.0 (18.97)
  SBP; Week 12; n=8, 8: number analyzed (Participants) | 8 | 8
  SBP; Week 12; n=8, 8 | 4.1 (13.17) | 7.1 (18.74)
  SBP; Week 24; n=9, 8 | 2.7 (17.00) | 6.1 (14.97)
  DBP; Week 0 (post-dose); n=9, 8 | 0.1 (5.40) | 0.6 (7.15)
  DBP; Week 4 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  DBP; Week 4 (pre-dose); n=8, 8 | -3.1 (3.72) | 1.0 (14.11)
  DBP; Week 4 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  DBP; Week 4 (post-dose); n=8, 8 | -4.8 (4.92) | 1.3 (12.90)
  DBP; Week 8 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  DBP; Week 8 (pre-dose); n=8, 8 | -7.8 (8.31) | 0.6 (14.23)
  DBP; Week 8 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  DBP; Week 8 (post-dose); n=8, 8 | -11.3 (9.92) | -1.0 (13.63)
  DBP; Week 12; n=8, 8: number analyzed (Participants) | 8 | 8
  DBP; Week 12; n=8, 8 | -2.9 (4.49) | 2.6 (12.34)
  DBP; Week 24; n=9, 8 | -5.2 (6.98) | 3.0 (14.93)

18. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the supine position after five minutes of rest for the participant. Baseline is the most recent recorded value before dosing on Day 1 (Week 0). Change from Baseline is calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Week 0 (post-dose), Weeks 4 and 8 (pre-dose and post-dose) Weeks 12 and 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Beats per minute
  Week 0 (post-dose); n=9, 8 | -0.8 (7.63) | -2.5 (5.37)
  Week 4 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4 (pre-dose); n=8, 8 | 0.8 (9.60) | -1.8 (8.17)
  Week 4 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 4 (post-dose); n=8, 8 | -6.8 (9.04) | -1.0 (9.80)
  Week 8 (pre-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8 (pre-dose); n=8, 8 | 0.0 (8.26) | -1.5 (6.55)
  Week 8 (post-dose); n=8, 8: number analyzed (Participants) | 8 | 8
  Week 8 (post-dose); n=8, 8 | -6.3 (6.39) | -2.1 (6.22)
  Week 12; n=8, 8: number analyzed (Participants) | 8 | 8
  Week 12; n=8, 8 | 1.6 (3.66) | -4.1 (6.64)
  Week 24; n=9, 8 | 2.2 (6.69) | -0.4 (6.99)

19. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained using a standardized ECG machine that measured heart rate, PR, QRS, QT and corrected QT interval (QTc). ECG measurements were done with the participant in a supine position having rested in this position for approximately 5 minutes before each reading. Clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings at worst-case post-Baseline are presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for worst-case post-Baseline is presented.
Time Frame: Up to Week 12
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Participants
  NCS | 6 | 6
  CS | 1 | 0

20. Secondary Outcome: Number of Participants With Abnormal 24-hour Holter Findings
Description: A Holter monitor is a type of continuous ambulatory ECG device used for quantitative assessment of abnormal rhythm events. Number of participants with abnormal 24-hour Holter findings is presented. Data was summarized for participants with at least 16 hours of data.
Time Frame: Week 0
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 9 | 8
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the start of study treatment up to Week 24
Description: AEs and SAEs were collected in the Safety Population which comprised of all randomized participants who took at least 1 dose of study treatment.
Arm/Group | Placebo | GSK3772847
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/8
Other Adverse Events (participants affected / at risk) | 7/9 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | GSK3772847 (N=8)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | GSK3772847 (N=8)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03393806/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT03393806/SAP_001.pdf